CLINICAL TRIAL: NCT01169246
Title: Efficacy of the ATP Switch Automatic Programming in ICD and CRT-D Implanted Patients
Brief Title: Efficacy of the ATP Switch Automatic Programming in Implantable Cardioverter Defibrillator (ICD) and Cardiac Resynchronization Therapy Defibrillator (CRT-D) Implanted Patients
Acronym: ASAP
Status: Terminated | Type: Observational
Why Stopped: Low recruitement rate
Sponsor: MicroPort CRM (Industry)
Collaborators: Sorin Group France SAS (Unknown)
Responsible Party: Sponsor
Other Study IDs: RTGX02-ASAP; RTGX02
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2015-02

CONDITIONS: Ventricular Arrythmias
Keywords: ATP,CRT, ICD PARADYM

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Paradym VR, DR and CRT models

SUMMARY:
Primary objective is to assess the efficacy of the new ATP Autoswitch function in simple, dual or triple chamber ICD.

DETAILED DESCRIPTION:
The efficacy rate of the ATP Auto-switch function, defined as the % of VT episodes successfully reduced, will be compared with 85%.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been implanted (primo implantation or replacement) with an ICD model PARADYM VR 8250, DR 8550, CRT 8750, CRT 8770 models or any similar or higher range device
* ATP Auto-switch function is programmed ON

Exclusion Criteria:

* Presence of a contra-indication to the ICD therapy
* Life expectancy less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICD/CRT-D implanted patients population
Sampling Method: Non-Probability Sample
Enrollment: 1254 (Actual)
Dates: Start 2009-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Ventricular Tachyarrhythmia episode | 2 years
  % of VT episode successfully reduced by the ATP Auto-switch

SECONDARY OUTCOMES:
Arrhythmia incidence | 2 years
  DEvice based data

CONTACTS AND LOCATIONS:
Overall Officials: SAVOURE Arnaud, MD, Principal Investigator — CHU Rouen
Locations (1):
- CHU Brest, Brest, France